CLINICAL TRIAL: NCT00366275
Title: Phase II of Immunochemotherapy, in Vivo Purging, PBSC Mobilization and Autotransplant in Patients With Relapsed or Refractory Follicular Lymphoma
Brief Title: Immunochemotherapy, in Vivo Purging, PBSC Mobilization and Autotransplant in Relapsed or Refractory Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Luca Arcaini, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML17165; LNH 1-02 (Other: IRCCS Policlinico San Matteo)
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Results first posted 2010-10-18 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Follicular Lymphoma
Keywords: follicular lymphoma; rituximab; immunochemotherapy; peripheral blood stem cells (PBSC) mobilization; in vivo purging; autotransplant; bcl-2 rearrangement; molecular response
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- In vivo purging autotransplant (Experimental)
  Interventions: Procedure: Immunochemotherapy, in vivo purging and autrotransplant

INTERVENTIONS:
Procedure: Immunochemotherapy, in vivo purging and autrotransplant — 2-4 courses every 3 weeks with rituximab 375 mg/m^2 on day 1, vincristine 1.4 mg/m^2 on day 2 and cyclophosphamide 400 mg/m^2 on days 2-6. Courses were started if granulocytes >1.5 · 10^9/l. The phase of peripheral blood stem cells (PBSC) mobilization coupled rituximab 375 mg/m^2 on days 1 and 9 with high-dose cytarabine (AraC) 2 g/m^2 every 12 hours on days 2 and 3. Granulocyte colony-stimulating factor (G-CSF)(5 mcg/kg/day subcutaneously) was administered from day 6. High-dose chemotherapy with autotransplant consisted of BEAM [carmustine (BCNU), etoposide, Cytarabine (AraC), melphalan] followed by the infusion of in vivo purged peripheral blood stem cells (PBSC) + 2 consolidation doses of rituximab 375 mg/m^2 on days +14 and +21 after autotransplant.

SUMMARY:
The purpose of this study is to determine the rate and duration of complete remission and molecular response in patients with relapsed/refractory follicular lymphoma, using a combined treatment with rituximab plus chemotherapy followed by in vivo purged peripheral blood stem cells (PBSC) mobilization and autotransplant.

DETAILED DESCRIPTION:
Autologous stem cell transplantation has been shown effective in the long-term control of follicular lymphoma. Lymphoma, however, can progress after high-dose treatments. Lymphoma cells have been proved to contaminate bone marrow and peripheral blood stem cells (PBSC) collections and may contribute to relapse after autotransplant. The presence in peripheral blood and marrow of PCR-detectable cells bearing the bcl-2 rearrangement appeared to be a surrogate marker of disease and the achievement of a bcl-2 negative status is associated with a lower risk of recurrence. Several methods have been attempted to abolish graft contamination: in vitro treatment with cytotoxic agents, in vitro treatment with anti-B-cell monoclonal antibodies and complement, immunomagnetic beads, positive selection of CD34+ cells. All these techniques usually produce loss of cells, are time-consuming and expensive, and neoplastic depletion is often partial with residual polymerase chain reaction (PCR)-positive cells in the graft.

In the last years the chimeric anti-CD20 monoclonal antibody Rituximab has been shown to be an effective therapeutic option for low-grade lymphoma. Owing to the different mechanism of action, the synergism with cytotoxic agents, and the non-overlapping toxicity, Rituximab is an ideal drug for combination with chemotherapy. On this basis, Rituximab has been used during mobilisation procedures as a tool to obtain in vivo purging and collection of lymphoma-free progenitor cells. In addition, several studies have demonstrated that the efficiency of peripheral blood stem cells (PBSC) harvested is not adversely affected by Rituximab and that engraftment and all parameters of hematopoietic recovery are not compromised. The incorporation of Rituximab into sequential high-dose therapy programs produced high rates of clinical and molecular remission in patients with indolent lymphoma, indicating that the antibody has an additive effect on chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory follicular lymphoma after chemotherapy
* Patients with relapsed or refractory follicular lymphoma after rituximab as single agent or with chemotherapy
* Patients with transformed follicular lymphoma
* CD20-positivity
* Age between 18 and 60 years
* Advanced Ann Arbor stage
* Normal cardiac, renal and hepatic functions
* Negativity for human immunodeficiency virus (HIV), hepatitis B virus (HBV) and hepatitis C virus (HCV)
* Total amount of anthracycline previously received < 300 mg/m^2

Exclusion criteria:

* Creatinine > 2 mg/dl
* Alanine transaminase (ALT) and alkaline phosphatase > 2N
* Cardiac or pulmonary disease
* Severe organic or psychiatric disease
* Positivity for human immunodeficiency virus (HIV), hepatitis B virus (HBV) and hepatitis C virus (HCV)
* Pregnancy, breastfeeding
* Cancer diagnosis in the 5 years before lymphoma diagnosis, except of non-melanoma skin cancer and Cervical Intraepithelial Neoplasia (CIN)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2002-01; Primary Completion 2007-01 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Lazzarino, M.D., Principal Investigator — Division of Hematology, IRCCS Policlinico S. Matteo, University of Pavia
Locations (1):
- Division of Hematology, IRCCS Policlinico S. Matteo, University of Pavia, Pavia, Italy

REFERENCES:
- [Background] Lazzarino M, Arcaini L, Bernasconi P, Alessandrino EP, Gargantini L, Cairoli R, Orlandi E, Astori C, Brusamolino E, Pagnucco G, Colombo AA, Calatroni S, Iacona I, Regazzi MB, Morra E. A sequence of immuno-chemotherapy with Rituximab, mobilization of in vivo purged stem cells, high-dose chemotherapy and autotransplant is an effective and non-toxic treatment for advanced follicular and mantle cell lymphoma. Br J Haematol. 2002 Jan;116(1):229-35. doi: 10.1046/j.1365-2141.2002.03256.x. PMID 11841421
- [Background] Arcaini L, Orlandi E, Alessandrino EP, Iacona I, Brusamolino E, Bonfichi M, Bernasconi P, Calatroni S, Tenore A, Montanari F, Troletti D, Pascutto C, Regazzi M, Lazzarino M. A model of in vivo purging with Rituximab and high-dose AraC in follicular and mantle cell lymphoma. Bone Marrow Transplant. 2004 Jul;34(2):175-9. doi: 10.1038/sj.bmt.1704551. PMID 15170171
- [Result] Arcaini L, Montanari F, Alessandrino EP, Tucci A, Brusamolino E, Gargantini L, Cairoli R, Bernasconi P, Passamonti F, Bonfichi M, Zoli V, Bottelli C, Calatroni S, Troletti D, Merli M, Pascutto C, Majolino I, Rossi G, Morra E, Lazzarino M. Immunochemotherapy with in vivo purging and autotransplant induces long clinical and molecular remission in advanced relapsed and refractory follicular lymphoma. Ann Oncol. 2008 Jul;19(7):1331-1335. doi: 10.1093/annonc/mdn044. Epub 2008 Mar 15. PMID 18344536
- [Derived] Arcaini L, Morello L, Tucci A, Rusconi C, Ladetto M, Rattotti S, Bonfichi M, Bottelli C, Gabutti C, Bernasconi P, Varettoni M, Gotti M, Troletti D, Guerrera ML, Fiaccadori V, Sciarra R, Ferretti VV, Alessandrino EP, Rossi G, Morra E. Autologous stem cell transplantation with in vivo purged progenitor cells shows long-term efficacy in relapsed/refractory follicular lymphoma. Am J Hematol. 2015 Mar;90(3):230-4. doi: 10.1002/ajh.23919. PMID 25502635

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2002 and September 2007, 64 patients with relapsed or refractory follicular lymphoma were enrolled in the trial
Groups:
- Immunochemotherapy, in Vivo Purging and Autotransplant: 2-4 courses every 3 weeks with rituximab 375 mg/m^2 on day 1, vincristine 1.4 mg/m^2 on day 2 and cyclophosphamide 400 mg/m^2 on days 2-6. Courses were started if granulocytes >1.5 · 109/l. The phase of peripheral blood stem cells (PBSC) mobilization coupled rituximab 375 mg/m^2 on days 1 and 9 with high-dose cytarabine (AraC) 2 g/m^2 every 12 hours on days 2 and 3. Granulocyte colony-stimulating factor (G-CSF)(5 mcg/kg/day s.c.) was administered from day 6. High-dose chemotherapy with autotransplant consisted of BEAM [carmustine (BCNU), etoposide, Cytarabine (AraC), melphalan] followed by the infusion of in vivo purged peripheral blood stem cells (PBSC) + 2 consolidation doses of rituximab 375 mg/m^2 on days +14 and +21 after autotransplant.
Period: Overall Study
Arm/Group | Immunochemotherapy, in Vivo Purging and Autotransplant
Started | 64
Completed | 58
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Immunochemotherapy, in Vivo Purging and Autotransplant
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 64
  >=65 years | 0
Age Continuous [Median (Full Range); unit: years] | 50 [44 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 35
Region of Enrollment [Number; unit: participants]
  Italy | 64

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: PFS is calculated according to the Kaplan-Meier estimator. The observation time of each subject is defined as the time from entry into the study until lymphoma progression or death as a result of any cause whichever occurs first.
  The 5-year PFS is the estimated cumulative probability of surviving at least 5 years without progression.
Time Frame: every 3 months for the first year after autotransplant and every 6 months after the first year of follow up
Measure: Number (95% Confidence Interval); unit: percent chance of PFS at 5 years
Arm/Group | Immunochemotherapy, in Vivo Purging and Autotransplant
Number analyzed (Participants) | 58
percent chance of PFS at 5 years | 59 [44 to 73]

ADVERSE EVENTS:
Arm/Group | Immunochemotherapy, in Vivo Purging and Autotransplant
Serious Adverse Events (participants affected / at risk) | 2/64
Other Adverse Events (participants affected / at risk) | 54/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunochemotherapy, in Vivo Purging and Autotransplant (N=64)
sepsis (General disorders) | 1 (64) — One patient developed Escherichia coli sepsis during cytopenia, did not harvest PBSC and required intensive support and i.v. antimicrobial therapy
Vasculitis (Vascular disorders) | 1 (64) — One patient developed vasculitis during the cytopenic phase after autotransplant that resolved completely with steroids.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunochemotherapy, in Vivo Purging and Autotransplant (N=64)
Hematological toxicity grade 3-4 (Blood and lymphatic system disorders) | 54 (64) — 44 patients out of 61 developed grade 3-4 hematological toxicity after high dose Ara-C while 10 aut of 59 developed grade 3-4 hematological toxicity during autotransplant

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes